CLINICAL TRIAL: NCT03828812
Title: Temporal Patterns of Diet and the Changes in Body Composition and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Hsin-Jen Chen, Assistant Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YM104136E
Record Dates: First submitted 2019-01-30; First posted 2019-02-04 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Body Composition; Blood Pressure; Mealtimes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breakfast promotion (Active Comparator): Receiving the recommendation of daily breakfast
  Interventions: Behavioral: Breakfast promotion
- Nighttime snack reduction (Active Comparator): Receiving the recommendation of reducing nighttime snack frequency
  Interventions: Behavioral: Nighttime snack reduction
- Breakfast promotion + nighttime snack reduction (Experimental): Receiving the recommendation of daily breakfast + reducing nighttime snack frequency
  Interventions: Behavioral: Breakfast promotion; Behavioral: Nighttime snack reduction

INTERVENTIONS:
Behavioral: Breakfast promotion — Recommendation of having breakfast daily
  Arms: Breakfast promotion; Breakfast promotion + nighttime snack reduction
Behavioral: Nighttime snack reduction — Recommendation of reducing frequency of nighttime snacking
  Arms: Breakfast promotion + nighttime snack reduction; Nighttime snack reduction

SUMMARY:
The study includes two parts: 1) an observational study examines the association of meal frequency, meal timing, and meal regularity with short-term changes in blood pressure and body composition; 2) a randomized controlled intervention examines the influence of recommendation of increase breakfast frequency and decrease nighttime snacking on 1-year changes in blood pressure and body composition.

ELIGIBILITY:
Inclusion criteria:

* Adult
* Willing to participate

Exclusion criteria:

* Being pregnant
* hemodialysis patients
* clinical diagnosis of cardiovascular diseases
* clinical diagnosis of cancer
* clinical diagnosis of dementia
* clinical diagnosis of eating disorders
* having metal orthopedic implants
* having pacemaker implanted

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Body weight | 1 year
  Body weight in kilogram
Standing height | 1 year
  Height in meters
Body fat% | 1 year
  Bioimpedance method (TANITA BC-418)
Body mass index | 1 year
  Weight and height will be combined to report BMI in kg/m^2
Systolic blood pressure | 1 year
  Measured in mmHg (Microlife BP 3MS1-4K)
Diastolic blood pressure | 1 year
  Measured in mmHg (Microlife BP 3MS1-4K)

SECONDARY OUTCOMES:
Frequency of breakfast per week | 1 year
  Self-report food frequency questionnaire(0-7 days/week)
Frequency of nighttime snacking per week | 1 year
  Self-report food frequency questionnaire(0-7 days/week)

OTHER OUTCOMES:
Sleep quality score | 1 year
  Pittsburgh Sleep Questionnaire(0-21 points): The higher scores, the worse sleep quality
Mood status | 1 year
  Depression, Anxiety, Stress Scale (DASS): The higher scores, the worse moods

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Jen Chen, PhD, Principal Investigator — National Yang Ming Chiao Tung University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen HJ, Tsai YC, Hsu YT, Chu J. Effect of recommendations of breakfast and late-evening snack habits on body composition and blood pressure: A pilot randomized trial. Chronobiol Int. 2024 Jul;41(7):1021-1033. doi: 10.1080/07420528.2024.2363492. Epub 2024 Jun 11. PMID 38860554